CLINICAL TRIAL: NCT04629469
Title: Low Field and High Field Magnetic Resonance Imaging Assessments on Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001356
Record Dates: First submitted 2020-10-27; First posted 2020-11-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Conditions Requiring a Brain Magnetic Resonance Imaging, Head Computerized Tomography, or Head Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hyperfine (Experimental): For patients that have standard of care head imaging, we will do a secondary analysis to compare their standard of care MRI, CT and/or US exams with Hyperfine MRI exams.
  Interventions: Diagnostic Test: Hyperfine MRI

INTERVENTIONS:
Diagnostic Test: Hyperfine MRI — • Patients who have a standard of care MRI, CT or US will undergo a low-field MRI utilizing Hyperfine either at the patient's bedside or in the department of Radiology. Results of the Hyperfine MRI will not be used for clinical care and will only be available to members of the research team for review.

SUMMARY:
Hyperfine Research, Inc. has taken advantage of technological advances and developed an MRI device that is not only portable, but also uses a very-low magnetic field strength, [less than 0.2 Tesla or approximately 10 times less] than the field strength of conventional devices. This critical difference allows HRI to address MRI's core challenges by, first, operating at very low magnetic field strengths, eliminating the need for special rooms or shielding. Second, there are minimal safety concerns regarding ferrous metals near the system, as the field strength is too low to attract metal objects. The removal of metal, including items such as jewelry, belts, etc. from clothing and person, prior to being scanned, is unnecessary. Third, the design constraints faced by conventional MRI systems are lifted at low magnetic field and an open device has been designed to minimize anxiety that may come with claustrophobic patients. All of this is possible while still providing image quality that is clinically relevant to a wide variety of fields, including radiology, neurology, pediatrics, emergency medicine, and others.

ELIGIBILITY:
Inclusion Criteria

Inpatients at CMH Adele Hall ages 0 days to 22 years are eligible for enrollment.

Exclusion Criteria

No additional sedation will be given as part of this study and that sedation, if already administered, will not be altered for study purposes.

Any patient who has a contraindication to having an MRI, such as:

Non-MRI conditional implanted device or device that is not able to be removed for MRI examination

Ages: 0 Days to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of hyperfine MRI versus conventional MRI, CT and/or US | Through study completion, an average of one year
  Sensitivity and specificity of hyperfine MRI versus conventional MRI, CT and/or US

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Chan, MD,PHD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sien ME, Robinson AL, Hu HH, Nitkin CR, Hall AS, Files MG, Artz NS, Pitts JT, Chan SS. Feasibility of and experience using a portable MRI scanner in the neonatal intensive care unit. Arch Dis Child Fetal Neonatal Ed. 2023 Jan;108(1):45-50. doi: 10.1136/archdischild-2022-324200. Epub 2022 Jul 4. PMID 35788031